CLINICAL TRIAL: NCT02123615
Title: ASIS for GAMMAGARD in Primary Immunodeficiency
Acronym: ASISinPI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ASIS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCTEB017805; 1R01EB017805 (Other Grant/Funding Number: NATIONAL INSTITUTE OF ALLERGY AND INFECTIOUS DISEASES)
Record Dates: First submitted 2014-04-11; First posted 2014-04-25 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Primary Immunodeficiency
Keywords: Primary Immunodeficiency; Subdermal bloodless space; Subdermal injection; Subcutaneous injection; Injectable electromyography needle; Electrical stimulation; MRI with Gadolinium
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Gadolinium; Gadolinium DTPA; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (20):
- Gadolinium For abdomen (Experimental): Gadolinium For abdomen Total Persistent % subdermally, For abdomen Total Persistent % subcutaneously, and For abdomen Relative Prolongation Ability Score.
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  1cc/ diluted with 19cc normal saline (for <40kg) or 29cc normal saline (for >40kg), subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium For abdomen; Drug: Gadolinium For lower back
- Gadolinium For lower back (Experimental): 1cc/ diluted with 19cc normal saline (for <40kg) or 29cc normal saline (for >40kg), subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Gadolinium For lower back Total Persistent % subdermally, For lower back Total Persistent % subcutaneously, and For lower back Relative Prolongation Ability Score.
  Interventions: Drug: Gadolinium For abdomen; Drug: Gadolinium For lower back
- subjects (%) of any infections (Experimental): subjects (%) of any infections as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- Annual rate of any infections (Experimental): Annual rate of any infections as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- subjects (%) with Antibiotic use (Experimental): subjects (%) with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- Annual rate with Antibiotic use (Experimental): Annual rate with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- subjects (%) with Days out of work (Experimental): subjects (%) with Days out of work as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- Annual rate with Days out of work (Experimental): Annual rate with Days out of work as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- (%) with hospitalized infections (Experimental): (%) with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- Annual rate hospitalized infections (Experimental): Annual rate hospitalized infections as Efficacy of Gammagard subcutaneously at Week 12, Efficacy of Gammagard subcutaneously at Week 24, and Efficacy of Gammagard subcutaneously at Week 36, vs. Efficacy of Gammagard subdermally at Week 12, Efficacy of Gammagard subdermally at Week 24, and Efficacy of Gammagard subdermally at Week 36.
  Interventions: Drug: Efficacy of Gammagard subcutaneously at Week 12; Drug: Efficacy of Gammagard subcutaneously at Week 24; Drug: Efficacy of Gammagard subcutaneously at Week 36; Drug: Efficacy of Gammagard subdermally at Week 36; Drug: Efficacy of Gammagard subdermally at Week 12; Drug: Efficacy of Gammagard subdermally at Week 24
- Adverse Injection Local Reactions (Experimental): Adverse Injection Local Reactions as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Headache (Experimental): Headache as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Fever (Experimental): Fever as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Nausea (Experimental): Nausea as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Vomiting (Experimental): Vomiting as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Fatigue (Experimental): Fatigue as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Diarrhea (Experimental): Diarrhea as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Asthma (Experimental): Asthma as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Oropharyngeal (Experimental): Oropharyngeal as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36
- Adverse Reactions Abdominal Pain (Experimental): Abdominal Pain as Adverse Reactions of Gammagard subcutaneously at Week 12, Adverse Reactions of Gammagard subcutaneously at Week 24, and Adverse Reactions of Gammagard subcutaneously at Week 36, vs. Adverse Reactions of Gammagard subdermally at Week 12, Adverse Reactions of Gammagard subdermally at Week 24, and Adverse Reactions of Gammagard subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Gammagard subcutaneously at Week 12; Drug: Adverse Reactions of Gammagard subcutaneously at Week 24; Drug: Adverse Reactions of Gammagard subcutaneously at Week 36; Drug: Adverse Reactions of Gammagard subdermally at Week 12; Drug: Adverse Reactions of Gammagard subdermally at Week 24; Drug: Adverse Reactions of Gammagard subdermally at Week 36

INTERVENTIONS:
Drug: Gadolinium For abdomen — Gadolinium 1cc/ diluted with 19cc normal saline (for <40kg) or 29cc normal saline (for >40kg) subdermally with ASIS Device for 30 patients.
  Gadolinium For abdomen Total Persistent % subdermally on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Gadolinium For abdomen; Gadolinium For lower back
Drug: Gadolinium For abdomen — Gadolinium 1cc/ diluted with 19cc normal saline (for <40kg) or 29cc normal saline (for >40kg) subcutaneously for 30 patients.
  Gadolinium For abdomen Total Persistent % subcutaneously on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Gadolinium For abdomen; Gadolinium For lower back
Drug: Gadolinium For abdomen — Gadolinium For abdomen Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium subcutaneously on MRI.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Gadolinium For abdomen; Gadolinium For lower back
Drug: Gadolinium For lower back — Gadolinium For lower back Total Persistent % subdermally on MRI at 6 hrs, 12 hrs, and 24 hrs. Gadolinium 1cc/ diluted with 19cc normal saline (for <40kg) or 29cc normal saline (for >40kg) subdermally with ASIS Device for 30 patients.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Gadolinium For abdomen; Gadolinium For lower back
Drug: Gadolinium For lower back — Gadolinium For lower back Total cumulative Persistent % of Gadolinium subcutaneously on MRI at 6 hrs, 12 hrs, and 24 hrs. Gadolinium 1cc/ diluted with 19cc normal saline (for <40kg) or 29cc normal saline (for >40kg) subcutaneously for 30 patients.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Gadolinium For abdomen; Gadolinium For lower back
Drug: Gadolinium For lower back — Gadolinium For lower back Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium subcutaneously on MRI .
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Gadolinium For abdomen; Gadolinium For lower back
Drug: Efficacy of Gammagard subcutaneously at Week 12 — subjects (%) of any infections as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — Annual rate of any infections as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — subjects (%) with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — Annual rate with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — subjects (%) with Days out of work as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — Annual rate with Days out of work as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — (%) with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 12 — Annual rate with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — subjects (%) of any infections as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — Annual rate of any infections as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — subjects (%) with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — Annual rate with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — subjects (%) with Days out of work as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — Annual rate with Days out of work as Efficacy of Gammagard subcutaneously at Week 24
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — (%) with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 24 — Annual rate with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 36 — subjects (%) of any infections as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 36 — Annual rate of any infections as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 36 — subjects (%) with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 36 — Annual rate with Antibiotic use as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subcutaneously at Week 36 — subjects (%) with Days out of work as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — Annual rate with Days out of work as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — (%) with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — Annual rate with hospitalized infections as Efficacy of Gammagard subcutaneously at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — subjects (%) of any infections as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — Annual rate of any infections as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — subjects (%) with Antibiotic use as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — Annual rate with Antibiotic use as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — subjects (%) with Days out of work as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — Annual rate with Days out of work as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — (%) with hospitalized infections as Efficacy of Gammagard subdermally at Week 12
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 12 — Annual rate with hospitalized infections as Efficacy of Gammagard subdermally at Week 12.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — subjects (%) of any infections as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — Annual rate of any infections as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — subjects (%) with Antibiotic use as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — Annual rate with Antibiotic use as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — subjects (%) with Days out of work as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — Annual rate with Days out of work as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — (%) with hospitalized infections as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 24 — Annual rate with hospitalized infections as Efficacy of Gammagard subdermally at Week 24.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — subjects (%) of any infections as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — Annual rate of any infections as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — subjects (%) with Antibiotic use as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — Annual rate with Antibiotic use as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — subjects (%) with Days out of work as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — Annual rate with Days out of work as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — (%) with hospitalized infections as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Efficacy of Gammagard subdermally at Week 36 — Annual rate with hospitalized infections as Efficacy of Gammagard subdermally at Week 36.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: (%) with hospitalized infections; Annual rate hospitalized infections; Annual rate of any infections; Annual rate with Antibiotic use; Annual rate with Days out of work; subjects (%) of any infections; subjects (%) with Antibiotic use; subjects (%) with Days out of work
Drug: Adverse Reactions of Gammagard subcutaneously at Week 12 — Adverse Reactions of Gammagard subcutaneously at Week 12, in number of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: Adverse Injection Local Reactions; Adverse Reactions Abdominal Pain; Adverse Reactions Asthma; Adverse Reactions Diarrhea; Adverse Reactions Fatigue; Adverse Reactions Fever; Adverse Reactions Headache; Adverse Reactions Nausea; Adverse Reactions Oropharyngeal; Adverse Reactions Vomiting
Drug: Adverse Reactions of Gammagard subcutaneously at Week 24 — Adverse Reactions of Gammagard subcutaneously at Week 24, in number of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: Adverse Injection Local Reactions; Adverse Reactions Abdominal Pain; Adverse Reactions Asthma; Adverse Reactions Diarrhea; Adverse Reactions Fatigue; Adverse Reactions Fever; Adverse Reactions Headache; Adverse Reactions Nausea; Adverse Reactions Oropharyngeal; Adverse Reactions Vomiting
Drug: Adverse Reactions of Gammagard subcutaneously at Week 36 — Adverse Reactions of Gammagard subcutaneously at Week 36, in number of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: Adverse Injection Local Reactions; Adverse Reactions Abdominal Pain; Adverse Reactions Asthma; Adverse Reactions Diarrhea; Adverse Reactions Fatigue; Adverse Reactions Fever; Adverse Reactions Headache; Adverse Reactions Nausea; Adverse Reactions Oropharyngeal; Adverse Reactions Vomiting
Drug: Adverse Reactions of Gammagard subdermally at Week 12 — Adverse Reactions of Gammagard subdermally at Week 12, in number of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: Adverse Injection Local Reactions; Adverse Reactions Abdominal Pain; Adverse Reactions Asthma; Adverse Reactions Diarrhea; Adverse Reactions Fatigue; Adverse Reactions Fever; Adverse Reactions Headache; Adverse Reactions Nausea; Adverse Reactions Oropharyngeal; Adverse Reactions Vomiting
Drug: Adverse Reactions of Gammagard subdermally at Week 24 — Adverse Reactions of Gammagard subdermally at Week 24, in number of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: Adverse Injection Local Reactions; Adverse Reactions Abdominal Pain; Adverse Reactions Asthma; Adverse Reactions Diarrhea; Adverse Reactions Fatigue; Adverse Reactions Fever; Adverse Reactions Headache; Adverse Reactions Nausea; Adverse Reactions Oropharyngeal; Adverse Reactions Vomiting
Drug: Adverse Reactions of Gammagard subdermally at Week 36 — Adverse Reactions of Gammagard subdermally at Week 36, in number of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain.
  Other Names: Gammagard [Immune Globulin Infusion (Human)]
  Arms: Adverse Injection Local Reactions; Adverse Reactions Abdominal Pain; Adverse Reactions Asthma; Adverse Reactions Diarrhea; Adverse Reactions Fatigue; Adverse Reactions Fever; Adverse Reactions Headache; Adverse Reactions Nausea; Adverse Reactions Oropharyngeal; Adverse Reactions Vomiting

SUMMARY:
ASIS Corporation (ASIS) has developed the only automatic injection system for delivery of injectable products to it's optimum/right spot, just outside of the fascia, which exists subdermally (between the skin and muscle). Bloodless basically implies longer lasting medicinal effects, and minimal side effects - advantages that reflect the NIH mission of enhancing health, lengthening life, and reducing the burdens of illness and disability. ASIS device is stabilized on the surface of the skin with negative pressure and emits an electrical current to create a bloodless cavity subdermally. ASIS device correctly, automatically, and consistently delivers therapeutic agents, yet requiring little skill of a practitioner - providing the steady and safe infusion into subdermal bloodless space of virtually any injectable product in addition to Botox, including GAMMAGARD LIQUID, Enbrel, Insulin, and Fillers, etc. According to the FDA, "This innovation will have major impact on the healthcare industry."

DETAILED DESCRIPTION:
Aim 1 would require 6 months, to demonstrate ASIS device's consistent performance on 60 subjects with Primary Immunodeficiency (PI), and the particular skin affected by this disease.

30 subjects will receive Gadolinium subcutaneously, and 30 subjects will receive Gadolinium subdermally with ASIS device. An MRI will be taken promptly after Gadolinium injection, as starting reference, to which subsequent MRI taken at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. Since there isn't a way to measure level of Gadolinium within it, or any other (e.g.

GAMMAGARD) for that matter, at least the Prolongation of Gadolinium may be approximated by the greater or longer Persistent % on MRI. However, this approximation can only work if the variables are minimized to the same population with Primary Immunodeficiency (PI), and the particular skin affected by it. Case in point, Primary Immunodeficiency (PI) patients are prone to infection, and tend to have scared skin with less vascularity, so expectantly will have prolonged Gadolinium subcutaneously Persistent %, which will be very different from the skin of normal patients, while the Gadolinium subdermally Persistent % may or may not change. Therefore, the Relative Prolongation Ability Score or total Persistent % subdermally over that of total Persistent % subcutaneously, will be different and very specific for the particular skin affected by Primary Immunodeficiency. However, they are valuable indicators that will help us modify the GAMMAGARD dosage and duration to inject into that "unknown" subdermal space for Aim 2.

Aim 2 would require 12 months, using GAMMAGARD, instead of Gadolinium, to demonstrate the advantages of ASIS device subdermally over subcutaneously, for the same Primary Immunodeficiency subjects. Of course that Relative Prolongation Ability Score in Aim1 will be valuable, but it isn't absolutely required to start Aim 2, because GAMMAGARD's Pharmacokinetics will be studied anyway, by following Peak and Trough levels of immunoglobulin G.

However, the Pharmacokinetics of subdermally injected GAMMAGARD will be just dependent on GAMMAGARD's diffusion out of that subdermal bloodless space; therefore, if GAMMAGARD getting into the bloodstream becomes so severely inhibited, then we can just change the osmolality of GAMMAGARD in the end. The therapeutic advantages of GAMMAGARD with ASIS device subdermally over subcutaneously will also be studied by comparing the reduction of Validated Acute Serious Bacterial Infections, adverse reactions, and injection site pain.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria in general and for Gadolinium:

  * Main Criteria for Inclusion: Eligible Ages: 12 Years to 65
  * Genders Eligible for Study: Both
  * Accepts Healthy Volunteers: Yes
  * Must be outpatient, male or female, of any race, between 18 and 65 years of age.
  * Must be able to understand the requirements of the study including maintaining a diary, and sign informed consent.
  * Must be in good general health as determined by investigator.
  * If female of childbearing potential, must have negative pregnancy test result at screening visit and practice reliable method of contraception
* Inclusion Criteria for Primary Immunodeficiency in particular:

  * Patients 12 years or older. This includes, but is not limited to, common variable immunodeficiency (CVID), X-linked agammaglobulinemia, congenital agammaglobulinemia, Wiskott-Aldrich syndrome, and severe combined immunodeficiencies1,2.

Exclusion Criteria:

* Exclusion Criteria for Primary Immunodeficiency in particular:

  * Females who are pregnant, nursing, or planning a pregnancy during the study period or who are not using a reliable means of contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Relative Prolongation Ability Score for Gadolinium subdermally injected | 6 months
  Gadolinium will be injected with ASIS subdermally (30) or conventional subcutaneous (30) for 60 adult subjects with Primary Immunodeficiency. The first MRI taken promptly after Gadolinium injection for each patient would be his or her reference of 100% Persistent, to which his or her subsequent MRI taken @ 6 hr, @ 12 hr, and @24hr later will be compared for Persistent %. This approximation can only work if the variables are minimized to the same population with Primary Immunodeficiency. The Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % subcutaneously, in Primary Immunodeficiency will be very valuable indicators for us to modify the GAMMAGARD dosage and duration for testing with that "unknown" subdermal bloodless space in Aim 2.

SECONDARY OUTCOMES:
Efficacy of GAMMAGARD subcutaneously vs. subdermally in Primary Immunodeficiency | 12 months
  The therapeutic efficacy of GAMMAGARD, in terms of reduction of Validated Acute Serious Bacterial Infections will be compared, eg. subjects (%) and Annual rate of any infections, subjects (%) and Annual rate of Antibiotic use, subjects (%) and Annual rate with Days out of work, subjects (%) and Annual rate of hospitalized infections, to demonstrate the advantages of ASIS device subdermally over subcutaneously for GAMMAGARD at Week 12, 24, and 36.

OTHER OUTCOMES:
Adverse Reactions of GAMMAGARD subcutaneously vs. subdermally in Primary Immunodeficiency | 12 months
  Adverse Reactions of GAMMAGARD, in numbers of Local Reactions, Headache, Fever, Nausea, Vomiting, Fatigue, Diarrhea, Asthma, Oropharyngeal, and Abdominal Pain will be compared, to demonstrate the advantages of ASIS device subdermally over subcutaneously for GAMMAGARD at Week 12, 24, and 36.

CONTACTS AND LOCATIONS:
Overall Officials: Li Nguyen, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM INC; Thanh Phung, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM, INC; Hanh Nguyen, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM,INC
Locations (1):
- Automatic Subdermal Injector System, Inc, Westminster, California, United States

REFERENCES:
- [Background] Paonessa DF, Goldstein JC. Anatomy and physiology of head and neck infections (with emphasis on the fascia of the face and neck). Otolaryngol Clin North Am. 1976 Oct;9(3):561-80. No abstract available. PMID 980495
- [Background] Magnevist (gadopentetate dimeglumine) Injection Product Information: http://pharma.bayer.com/scripts/pages/en/products/diagnostic_imaging/index.php
- [Background] Botox (onabotulinumtoxinA) Product Information: http://www.botoxcosmetic.com/botox_physician_info/Clinical_Information.aspx http://www.clinicaltrials.gov/ct2/show/NCT01313767?term=Botox+pi&rank=1
- [Background] GAMMAGARD LIQUID Comparison of Intravenous and Subcutaneous Administration in Primary Immunodeficiency Diseases (PID): http://www.clinicaltrials.gov/ct2/show/NCT00546871?term=Gammagard+subcutaneous&rank=5
- [Background] Daw Z, Padmore R, Neurath D, Cober N, Tokessy M, Desjardins D, Olberg B, Tinmouth A, Giulivi A. Hemolytic transfusion reactions after administration of intravenous immune (gamma) globulin: a case series analysis. Transfusion. 2008 Aug;48(8):1598-601. doi: 10.1111/j.1537-2995.2008.01721.x. Epub 2008 May 2. PMID 18466176
- [Background] Mignogna MD, Fortuna G, Ruoppo E, Adamo D, Leuci S, Fedele S. Variations in serum hemoglobin, albumin, and electrolytes in patients receiving intravenous immunoglobulin therapy: a real clinical threat? Am J Clin Dermatol. 2007;8(5):291-9. doi: 10.2165/00128071-200708050-00004. PMID 17902731
- [Background] Kreil TR, Berting A, Kistner O, Kindermann J. West Nile virus and the safety of plasma derivatives: verification of high safety margins, and the validity of predictions based on model virus data. Transfusion. 2003 Aug;43(8):1023-8. doi: 10.1046/j.1537-2995.2003.00496.x. PMID 12869106
- [Background] Ochs HD, Gupta S, Kiessling P, Nicolay U, Berger M; Subcutaneous IgG Study Group. Safety and efficacy of self-administered subcutaneous immunoglobulin in patients with primary immunodeficiency diseases. J Clin Immunol. 2006 May;26(3):265-73. doi: 10.1007/s10875-006-9021-7. PMID 16783465
- [Background] Gardulf A, Nicolay U, Asensio O, Bernatowska E, Bock A, Carvalho BC, Granert C, Haag S, Hernandez D, Kiessling P, Kus J, Pons J, Niehues T, Schmidt S, Schulze I, Borte M. Rapid subcutaneous IgG replacement therapy is effective and safe in children and adults with primary immunodeficiencies--a prospective, multi-national study. J Clin Immunol. 2006 Mar;26(2):177-85. doi: 10.1007/s10875-006-9002-x. Epub 2006 Apr 26. PMID 16758340
- [Background] Orange JS, Hossny EM, Weiler CR, Ballow M, Berger M, Bonilla FA, Buckley R, Chinen J, El-Gamal Y, Mazer BD, Nelson RP Jr, Patel DD, Secord E, Sorensen RU, Wasserman RL, Cunningham-Rundles C; Primary Immunodeficiency Committee of the American Academy of Allergy, Asthma and Immunology. Use of intravenous immunoglobulin in human disease: a review of evidence by members of the Primary Immunodeficiency Committee of the American Academy of Allergy, Asthma and Immunology. J Allergy Clin Immunol. 2006 Apr;117(4 Suppl):S525-53. doi: 10.1016/j.jaci.2006.01.015. PMID 16580469
- [Background] Bonilla FA, Bernstein IL, Khan DA, Ballas ZK, Chinen J, Frank MM, Kobrynski LJ, Levinson AI, Mazer B, Nelson RP Jr, Orange JS, Routes JM, Shearer WT, Sorensen RU; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. Practice parameter for the diagnosis and management of primary immunodeficiency. Ann Allergy Asthma Immunol. 2005 May;94(5 Suppl 1):S1-63. doi: 10.1016/s1081-1206(10)61142-8. No abstract available. PMID 15945566
- [Background] Kahwaji J, Barker E, Pepkowitz S, Klapper E, Villicana R, Peng A, Chang R, Jordan SC, Vo AA. Acute hemolysis after high-dose intravenous immunoglobulin therapy in highly HLA sensitized patients. Clin J Am Soc Nephrol. 2009 Dec;4(12):1993-7. doi: 10.2215/CJN.04540709. Epub 2009 Oct 15. PMID 19833910
- See also: Click here for more information about this study ASIS for GAMMAGARD in Primary Immunodeficiency — http://www.asis-inc.com